CLINICAL TRIAL: NCT04080752
Title: Double-Blind, Placebo-Controlled, Multi-Center Study Investigating the Efficacy, Safety, and Tolerability of JNJ-61393215 as Adjunctive Treatment in Adults With Major Depressive Disorder With Anxious Distress With Suboptimal Response to Standard Antidepressants
Brief Title: A Study of JNJ-61393215 in the Treatment of Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108655; 2019-001683-29 (EudraCT Number); 61393215MDD2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Results first posted 2022-09-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder With Anxious Distress
MeSH Terms: interventions — Hcrtr1 protein, mouse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JNJ-61393215 135 milligram (mg) (Experimental): Participants will receive JNJ-61393215 135 mg (3*45 mg capsules) orally once daily for 6 weeks along with the prescribed standard oral antidepressants (without dose change) throughout the study.
  Interventions: Drug: JNJ-61393215
- Placebo (Placebo Comparator): Participants will receive matching placebo for 6 weeks along with the prescribed standard oral antidepressants (without dose change) throughout the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-61393215 — JNJ-61393215 will be administrated orally.
  Other Names: Orexin-1
  Arms: JNJ-61393215 135 milligram (mg)
Drug: Placebo — Matching placebo will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of JNJ-61393215 as adjunctive treatment compared to adjunctive placebo, as assessed by the change from baseline to week 6 on a 17-item Hamilton Depression Rating Scale (HDRS-17) in participants with major depressive disorder (MDD) with anxious distress with a score greater than or equal to (>=) 2 on item 26 or 27 of the Inventory of Depressive Symptomatology, Clinician Rating -30 (IDS-C30), who have a suboptimal response to current treatment with a standard antidepressant.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a body mass index (BMI) between 18 and 36 kilogram per meter square (kg/m^2)
* Participants must have a primary diagnostic and statistical manual of mental disorders, 5th edition (DSM-5) diagnosis of major depressive disorder (MDD) with anxious distress, as assessed by the mini international neuropsychiatric inventory 7.0. Plus (MINI). Participants with a diagnosis of comorbid generalized anxiety disorder (GAD), post-traumatic stress disorder, persistent depressive disorder, attention deficit hyperactivity disorder (ADHD), social anxiety disorder or nicotine/caffeine dependence may be included, if MDD is primary diagnosis
* Participants must have an inventory of depressive symptomatology, clinician rating-30 (IDS-C30) total score greater than or equal to (>=) 35 (moderate to severe depression)
* Participant must not have received more than 3 failed antidepressant treatments (of adequate dose and duration), including their current treatment, in the current episode of depression, as documented by the massachusetts general hospital antidepressant treatment history questionnaire (MGH-ATRQ)
* Participant must be currently receiving 1 of the following antidepressants for at least 6 weeks duration at screening, at an adequate therapeutic dose, as determined by the MGH-ATRQ and should remain on a stable dose throughout the study: bupropion, citalopram, escitalopram, sertraline, paroxetine, venlafaxine, desvenlafaxine, duloxetine, fluoxetine, vilazodone, vortioxetine, mirtazapine, agomelatine, nortriptyline, imipramine, amitriptyline and levomilnacipran
* Participants must have a suboptimal response (improvement <50%) to the antidepressant used as their current treatment, as measured by the MGH-ATRQ
* A woman of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test before the first dose

Exclusion Criteria:

* Participant has any other psychiatric condition including but not limited to: MDD with current psychotic features, bipolar disorder (including lifetime diagnosis), obsessive-compulsive disorder, borderline personality disorder, eating disorder (example: bulimia, anorexia nervosa), or schizophrenia (lifetime)
* Age of onset of depression is after 55 years of age
* Participant has a history of alcohol or substance use disorder (abuse/dependence) within 6 months prior to screening (nicotine and caffeine dependence are not exclusionary)
* Participant has a current or recent (within the past year) history of clinically significant suicidal ideation (corresponding to a score of >= 3 for ideation) or any suicidal behavior within the past year, as validated on the Colombia suicide severity rating scale (C-SSRS) at screening or baseline
* Length of current major depressive episode >60 months
* Participant has organic brain disease or dementia or has known or suspected intellectual development disorder
* Participant has been treated with at least one of the following treatments: (a) electroconvulsive therapy in the current episode; (b) deep brain stimulation (lifetime); (c) repetitive transcranial magnetic stimulation within 4 weeks prior to baseline visit
* Participant has any clinically relevant medical condition that could potentially alter the absorption, metabolism, or excretion of the study intervention, such as liver disease or renal disease
* Participant has a relevant history of any significant and/or unstable cardiovascular, respiratory, neurological (including seizures - uncomplicated childhood febrile seizures with no sequelae are not exclusionary) or significant cerebrovascular, renal, hepatic, dermatologic, hematologic, gastrointestinal or endocrine diseases. Hospitalization for cardiovascular event (myocardial infarction, unstable angina, stroke, transient ischemic attack) within 3 months prior to the first administration of study drug is exclusionary. Diabetes mellitus be allowed when the participant is stable (HbA1c less than 7.5% or 58 mmol/mol)
* Participant has a clinically significant abnormal physical examination, vital signs or 12-lead electrocardiogram (ECG) at screening or baseline Minor deviations in ECG, which are not considered to be of clinical significance to the investigator, are acceptable.If at screening visit QTcB or QTcF interval >=450 ms for males or >=470 ms for females, or >480 ms if bundle branch block and prolongation of the QTc interval are present;participant is excluded
* Participant has a history of known demyelinating diseases such as multiple sclerosis or optic neuritis

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 222 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (35):
- United States (9):
  - Collaborative NeuroScience Network, Garden Grove, California
  - Atlanta Institute, Alpharetta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - The Medical Research Network, LLC, New York, New York
  - Richmond Behavioural Associates, Staten Island, New York
  - Ohio State University, Columbus, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
- ARENSIA, Chisinau, Moldova
- Russia (13):
  - City Clinical Psychiatric Hopsital 3, Moscow
  - Nizny Novgorod clinical psychiatric hospital 1, Nizny Novgorod
  - Orenburg Regional Clinical Psychiatric Hospital #1, Orenburg
  - Medical and Rehabilitation Research Center Phoenix, Rostov-on-Don
  - Psychoneurological dispensary 10, Saint Petersburg
  - City Psychiatric hospital 7 named after I.P.Pavlov, Saint Petersburg
  - Psychoneurological dispensary 1, Saint Petersburg
  - SHI 'Saratov City Clinical Hospital 2 n.a V.I. Razumovsky, Saratov
  - Saratov Regional Psychiatric hospital named after St. Sofia, Saratov
  - Engels psychiatric hospital, Saratov Region
  - Psychoneurological Dispensary #4, St.Peterburg
  - Stavropol Region Psychiatric Hospital #2, Stavropol
  - Research Institute of Mental Health, Tomsk
- Ukraine (8):
  - MNCE of Kyiv RC Regional Psychiatric and Narcological Medical Association, Hlevakha
  - CNCE'Precarpathian Regional Clinical Mental Health Center Ivano-Frankivsk RC', Ivano-Frankivsk
  - Mnpe of Kharkiv Regional Council 'Regional Clinical Psychiatric Hospital #3', Kharkiv
  - CNPE'Kherson Regional Institution of Mental Care'of Kherson Regional Council, Kherson
  - Kyiv Railway Station Clinical Hospital #2, Kyiv
  - Mnpe 'Regional Clinical Psychiatric Hospital of Kirovohrad Regional Council', Nove
  - CNCE 'Cherkasy Regional Psychiatric Hospital of Cherkasy Regional Council', Smila
  - CNCE 'Vinnytsya RC Psychoneurological Hospital n.a. O.I. Yushchenko Vinnytsya RC', Vinnytsia
- United Kingdom (4):
  - MAC Clinical Research, Barnsley
  - MAC Clinical Research, Liverpool
  - Kings College London, London
  - MAC Clinical Research, Manchester

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Schmidt ME, Moyer JA, Kezic I, Zhou X, Samtani MN, Bleys C, Dallas S, Salvadore G, Drevets WC. Efficacy, safety, and tolerability of JNJ-61393215 (tebideutorexant), a selective orexin-1 receptor antagonist, as adjunctive treatment for major depressive disorder with anxious distress: A double-blind, placebo-controlled, randomized phase 2a study. Eur Neuropsychopharmacol. 2025 Jun;95:14-23. doi: 10.1016/j.euroneuro.2025.03.007. Epub 2025 Apr 13. PMID 40215570

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: After a screening period of up to 4 weeks duration, participants received placebo matching to JNJ-61393215 capsule orally once daily during 6 weeks double-blind treatment period, followed by 2 weeks post treatment follow-up period. Throughout the study, participants continued their standard treatment of oral antidepressants at an adequate and tolerated stable dose.
- JNJ-61393215 135 Milligrams (mg): After a screening period of up to 4 weeks duration, participants received JNJ-61393215 135 mg (3*45 mg) capsule orally once daily during 6 weeks double-blind treatment period, followed by 2 weeks post treatment follow-up period. Throughout the study, participants continued their standard treatment of oral antidepressants at an adequate and tolerated stable dose.
Period: Overall Study
Arm/Group | Placebo | JNJ-61393215 135 Milligrams (mg)
Started | 112 | 110
Completed | 99 | 104
Not Completed | 13 | 6
Not completed — Adverse Event | 2 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Non-Compliance with Study Drug | 0 | 1
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all randomized participants who received at least 1 dose of study agent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | JNJ-61393215 135 Milligrams (mg) | Total
Number analyzed (Participants) | 112 | 110 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (12.99) | 43.6 (12.39) | 41.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 88 | 167
  Male | 33 | 22 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 13 | 26
  White | 97 | 95 | 192
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  MOLDOVA, REPUBLIC OF | 18 | 17 | 35
  RUSSIAN FEDERATION | 36 | 34 | 70
  UKRAINE | 22 | 21 | 43
  UNITED KINGDOM | 10 | 9 | 19
  UNITED STATES | 26 | 29 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Depression Rating Scale-17 (HDRS-17) Total Score at Week 6
Description: Change from baseline in HDRS-17 total score at Week 6 was reported. The HDRS-17 is a clinician-administered rating scale designed to assess the severity of symptoms in participants diagnosed with depression with a score range of 0 to 52. Each of the 17 items is rated by the clinician on either a 3-point (0 to 2) or a 5-point scale (0 to 4). The point scale used a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). A total score (range: 0 to 52) was calculated by adding the scores of all 17 items. For each item as well as the total score, a higher score represents a more severe condition (greater depression).
Time Frame: Baseline and Week 6
Population: The enriched analysis set (EAS) included all randomized participants who received at least 1 dose of study agent and had improvement in percent changes in HDRS17 total score less than (<)25 percent (%) from screening to baseline and HDRS-17 total score greater than or equal to (>=)18 at baseline. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | JNJ-61393215 135 Milligrams (mg)
Number analyzed (Participants) | 97 | 103
Units on a scale | -8.8 (0.66) | -9.4 (0.64)
Statistical Analysis 1: Comparison: Placebo vs JNJ-61393215 135 Milligrams (mg); Test type: Superiority; p = 0.2494, Mixed Model for Repeated Measures (MMRM); Least Square (LS) Mean Difference = -0.61, 80% CI 2-sided [-1.76 to 0.55], Standard Error of Mean 0.897

2. Secondary Outcome: Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score at Week 6
Description: Change from baseline in HAM-A total score at Week 6 was reported. HAM-A is a 14-item scale designed to measure severity of anxiety-related symptoms in participants. Each question reflects a symptom of general anxiety, including physical anxiety and mental anxiety. Each item was rated on a 5-point scale ranged from 0 (not present) to 4 (maximum anxiety). The total score was sum of 14 items scores and it ranged from 0 (normal) to 56 (severe), where higher score indicated greater degree of anxiety symptom. The total score was categorized as 0-13: normal range, 14-17: mild severity, 18-24: mild to moderate severity, 25-30: moderate to severe, and >=31: severe. Negative change in score indicates improvement.
Time Frame: Baseline and Week 6
Population: The EAS included all randomized participants who received at least 1 dose of study agent and had improvement in percent changes in HDRS17 total score <25% from screening to baseline and HDRS-17 total score >=18 at baseline. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | JNJ-61393215 135 Milligrams (mg)
Number analyzed (Participants) | 97 | 103
Units on a scale | -10.4 (0.74) | -10.3 (0.72)

3. Secondary Outcome: Change From Baseline in HAM-A Total Score at Weeks 2 and 4
Description: Change from baseline in HAM-A total score at Weeks 2 and 4 were reported. HAM-A is a 14-item scale designed to measure severity of anxiety-related symptoms in participants. Each question reflects a symptom of general anxiety, including physical anxiety and mental anxiety. Each item was rated on a 5-point scale ranged from 0 (not present) to 4 (maximum anxiety). The total score was sum of 14 items scores and it ranged from 0 (normal) to 56 (severe), where higher score indicated greater degree of anxiety symptom. The total score was categorized as 0-13: normal range, 14-17: mild severity, 18-24: mild to moderate severity, 25-30: moderate to severe, and >=31: severe. Negative change in score indicates improvement.
Time Frame: Baseline, Week 2, and Week 4
Population: The EAS included all randomized participants who received at least 1 dose of study agent and had improvement in percent changes in HDRS17 total score <25% from screening to baseline and HDRS-17 total score >=18 at baseline. Here, 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. Here, 'n' (number analyzed) signifies participants evaluable for this outcome measure at specified time points.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | JNJ-61393215 135 Milligrams (mg)
Number analyzed (Participants) | 105 | 108
Units on a scale
  Week 2 | -4.85 (0.511) | -4.1 (0.505)
  Week 4: number analyzed (Participants) | 99 | 105
  Week 4 | -8.05 (0.616) | -7.9 (0.603)

4. Secondary Outcome: Change From Baseline in HDRS-17 Total Score in Participants With a Baseline HAM-A Score >=20 at Week 6
Description: Change from baseline in HDRS-17 total score in participants with a baseline HAM-A score >=20 at Week 6 was reported. The HDRS-17 is a clinician-administered rating scale designed to assess the severity of symptoms in participants diagnosed with depression with a score range of 0 to 52. Each of the 17 items is rated by the clinician on either a 3-point (0 to 2) or a 5-point scale (0 to 4). The point scale used a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). A total score (range: 0 to 52) was calculated by adding the scores of all 17 items. For each item as well as the total score, a higher score represents a more severe condition (greater depression).
Time Frame: Baseline and Week 6
Population: The analyzed population included participants of EAS who had baseline HAM-A Score of >=20.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | JNJ-61393215 135 Milligrams (mg)
Number analyzed (Participants) | 91 | 94
Units on a scale | -8.8 (0.68) | -9.8 (0.67)

5. Secondary Outcome: Change From Baseline in HAM-A Total Score in Participants With a Baseline HAM-A Score >=20 at Week 6
Description: Change from baseline in HAM-A total score in participants with a baseline HAM-A score >=20 at Week 6 was reported. HAM-A is a 14-item scale designed to measure severity of anxiety-related symptoms in participants. Each question reflects a symptom of general anxiety, including physical anxiety and mental anxiety. Each item was rated on a 5-point scale ranged from 0 (not present) to 4 (maximum anxiety). The total score was sum of 14 items scores and it ranged from 0 (normal) to 56 (severe), where higher score indicated greater degree of anxiety symptom. The total score was categorized as 0-13: normal range, 14-17: mild severity, 18-24: mild to moderate severity, 25-30: moderate to severe, and >=31: severe. Negative change in score indicates improvement.
Time Frame: Baseline and Week 6
Population: The analyzed population included participants of EAS who had baseline HAM-A Score of >=20.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | JNJ-61393215 135 Milligrams (mg)
Number analyzed (Participants) | 91 | 94
Units on a scale | -10.6 (0.78) | -10.9 (0.77)

6. Secondary Outcome: Change From Baseline in Generalized Anxiety Disorder-7 (GAD-7) Total Score at Week 6
Description: Change from baseline in GAD-7 total score at Week 6 was reported. The GAD-7 is a brief and validated 7-item self-reported assessment of overall anxiety. Participants respond to each item using a 4-point scale with response categories of 0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day. Item responses are summed to yield a total score with a range of 0 to 21, where higher scores indicate more anxiety. The recall period is 2 weeks. The severity of the GAD-7 is categorized as follows: None (0-4), Mild (5-9), Moderate (10-14) and Severe (15-21).
Time Frame: Baseline and Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | JNJ-61393215 135 Milligrams (mg)
Number analyzed (Participants) | 97 | 102
Units on a scale | -5.3 (0.52) | -5.7 (0.51)

7. Secondary Outcome: Change From Baseline in Patient Health Questionnaire (PHQ-9) Total Score at Weeks 2 and 4
Description: Change From baseline in PHQ-9 total score at Weeks 2 and 4. The PHQ-9 is a 9-item, Patient Reported Outcome (PRO) measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) major depressive disorder (MDD) criteria. Each item is rated on a 4 point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participants item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms. The severity of the PHQ-9 is categorized as follows: None-minimal (0-4), Mild (5-9), Moderate (10-14), Moderately Severe (15-19) and Severe (20-27).
Time Frame: Baseline, Week 2, and Week 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | JNJ-61393215 135 Milligrams (mg)
Number analyzed (Participants) | 105 | 108
Units on a scale
  Week 2 | -3.26 (0.461) | -2.84 (0.455)
  Week 4: number analyzed (Participants) | 98 | 105
  Week 4 | -5.63 (0.557) | -5.71 (0.544)

8. Secondary Outcome: Change From Baseline in HDRS-17 Total Score at Weeks 2 and 4
Description: Change From baseline in HDRS-17 total score at Weeks 2 and 4. The HDRS-17 is a clinician-administered rating scale designed to assess the severity of symptoms in participants diagnosed with depression with a score range of 0 to 52. Each of the 17 items is rated by the clinician on either a 3-point (0 to 2) or a 5-point scale (0 to 4). The point scale used a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). A total score (range: 0 to 52) was calculated by adding the scores of all 17 items. For each item as well as the total score, a higher score represents a more severe condition (greater depression).
Time Frame: Baseline, Week 2, and Week 4
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | JNJ-61393215 135 Milligrams (mg)
Number analyzed (Participants) | 105 | 108
Units on a scale
  Week 2 | -3.98 (0.47) | -3.54 (0.465)
  Week 4: number analyzed (Participants) | 99 | 105
  Week 4 | -6.78 (0.546) | -7.03 (0.536)

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) as a Measure of Safety and Tolerability
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were events during the initiation of study drug up till follow-up period.
Time Frame: Up to 8 weeks
Population: The safety analysis set included all randomized participants who received at least 1 dose of study agent.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | JNJ-61393215 135 Milligrams (mg)
Number analyzed (Participants) | 112 | 110
Participants | 34 | 50

10. Secondary Outcome: Total Plasma Concentration of JNJ-61393215
Description: Total plasma concentration of JNJ-61393215 was reported. The concentrations of JNJ-61393215 were measured using a validated, specific, and sensitive liquid chromatography-mass spectrometry/mass spectrometry (LC-MS/MS) method.
Time Frame: 1-4 hours postdose on Day 1; Predose and 1-4 hours post dose on Days 15, 29, and 43
Population: Analysis population included participant who received JNJ-61393215 and for whom at least one pharmacokinetic (PK) concentration was available. Here, 'n' (number analyzed) signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: Nanograms per milliter (ng/mL)
Arm/Group | JNJ-61393215 135 Milligrams (mg)
Number analyzed (Participants) | 106
Nanograms per milliter (ng/mL)
  Day 1: 1-4 hours postdose: number analyzed (Participants) | 101
  Day 1: 1-4 hours postdose | 4143 (2315)
  Day 15: Predose: number analyzed (Participants) | 105
  Day 15: Predose | 3053 (1857)
  Day 15: 1-4 hours postdose: number analyzed (Participants) | 102
  Day 15: 1-4 hours postdose | 5638 (2362)
  Day 29: Predose | 3104 (1839)
  Day 29: 1-4 hours postdose: number analyzed (Participants) | 104
  Day 29: 1-4 hours postdose | 5868 (2267)
  Day 43: Predose: number analyzed (Participants) | 95
  Day 43: Predose | 3019 (1794)
  Day 43: 1-4 hours postdose: number analyzed (Participants) | 94
  Day 43: 1-4 hours postdose | 5897 (2288)

11. Secondary Outcome: Plasma Protein Binding (PPB): Percentage of JNJ-61393215 Unbound
Description: Percentage of JNJ-61393215 unbound was determined by using a liquid chromatography-mass spectrometry/mass spectrometry (LC-MS/MS) method. The protein binding was assessed by spiking plasma samples with radiolabeled JNJ-61393215.
Time Frame: Predose and 1-4 hours post dose on Day 43
Population: Analysis population included participant who received JNJ-61393215 and for whom PPB assessment was performed.
Measure: Mean (Standard Deviation); unit: Percentage of JNJ-61393215 unbound
Arm/Group | JNJ-61393215 135 Milligrams (mg)
Number analyzed (Participants) | 94
Percentage of JNJ-61393215 unbound
  Day 43: Predose | 2.52 (0.776)
  Day 43: 1-4 hours postdose | 4.15 (1.58)

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Description: The safety analysis set included all randomized participants who received at least 1 dose of study agent.
Arm/Group | Placebo | JNJ-61393215 135 Milligrams (mg)
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/110
Other Adverse Events (participants affected / at risk) | 12/112 | 30/110
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=112) | JNJ-61393215 135 Milligrams (mg) (N=110)
Abdominal Pain (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 1 | 6
Fatigue (General disorders) | 0 | 3
Urinary Tract Infection (Infections and infestations) | 0 | 3
Headache (Nervous system disorders) | 9 | 13
Somnolence (Nervous system disorders) | 0 | 9

LIMITATIONS AND CAVEATS:
The study was limited to a single dose level. During the study, the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic emerged. Public health measures required progressive restriction of movement of participants, site staff, and sponsor staff. The recruitment and enrollment were halted on 17 March 2020. All ongoing participants were permitted to continue the study if they were able to attend the on-site scheduled visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT04080752/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT04080752/SAP_001.pdf